CLINICAL TRIAL: NCT04195490
Title: Evaluation of the Outcomes of Feminizing Genitoplasty in Children With Disorders of Sex Development
Brief Title: Evaluation of Outcomes of Feminizing Genitoplasty in Children With Disorders of Sex Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hussein Ibrahim Ahmed, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: disorders of sex development
Record Dates: First submitted 2019-12-03; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Disorders of Sex Development
Keywords: feminizing genitoplasty
MeSH Terms: conditions — Disorders of Sex Development

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children with disorders of sex development (Other): children with disorders of sex development needing feminizing genitoplasty
  Interventions: Procedure: feminizing genitoplasty

INTERVENTIONS:
Procedure: feminizing genitoplasty — feminizing genitoplasty including vaginoplasty,clitroplasty, labioplasty and urethroplasty

SUMMARY:
Evaluate the short term outcomes of feminizing genitoplasty including vaginoplasty,clitroplasty, labioplasty and urethroplasty in children with disorders of sex development as regarding cosmetic and functional aspects.

DETAILED DESCRIPTION:
Disorders of sex development (DSD) are a wide range of congenital conditions characterized by incongruent development of the components involved in sex differentiation including chromosomes, gonads, brain and anatomic sex.Sex assignment is a critical aspect in management of DSD and it is determined by investigations, genital appearance, fertility potential and cultural practices and pressurs. It is recommended that genital surgery for a child raised as a female considered only in cases of severe virilization (Prader 3-5) and that surgery for the clitoris not be performed for reasons of cosmesis only.Feminizing genital reconstruction has evolved considerably over the past decades as a result of improved understanding of anatomy , modification of surgical procedures and audit of outcomes. For patients with congenital adrenal hyperplasia (CAH) with severe virilization raised as a female , it is recommended that clitorial and perineal reconstruction be considered in infancy and those with a low vaginal confluence undergo vaginoplasty at an early age , the appropriate timing for those with higher vaginal confluence is still less certain. Cosmetic outcomes after genitoplasty are variable. Most studies have detected only functional and cosmetic outcomes rated by the physician, but satisfaction ratings may differ between physicians and patients or their parents . The present prospective , interventional study aimed to describe the frequency of sex assignment and types of surgery performed in a cohort of patients with moderate to severe genital ambiguity and also evaluate surgical outcomes of feminizing genitoplasty in these patients .

ELIGIBILITY:
Inclusion Criteria:

1. Age : infants and children from 18 months old age to 14 years.
2. virilized external genitalia.

Exclusion Criteria:

* (1)children who did any corrective genitoplasty before. (2)children with debatable sex of rearing;ovotesticular DSD, mixed gonadal dysgenesis and partial androgen insensitivity.

Ages: 18 Months to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
The vaginal size will be evaluated for stenosis within 6 months after the procedure using Hegar dilators under general anaesthesia to ensure patency of the vagina. | 1 year
  The incidence of unsatisfied cosmetic results after feminizing genitoplasty

CONTACTS AND LOCATIONS:
Overall Officials: Hussein F Ibrahim, Msc, Principal Investigator — Assiut University; Tarek Sabra, MD, Study Director — Assiut University

REFERENCES:
- [Background] Lee PA, Houk CP, Ahmed SF, Hughes IA; International Consensus Conference on Intersex organized by the Lawson Wilkins Pediatric Endocrine Society and the European Society for Paediatric Endocrinology. Consensus statement on management of intersex disorders. International Consensus Conference on Intersex. Pediatrics. 2006 Aug;118(2):e488-500. doi: 10.1542/peds.2006-0738. No abstract available. PMID 16882788
- [Background] Sircili MH, e Silva FA, Costa EM, Brito VN, Arnhold IJ, Denes FT, Inacio M, de Mendonca BB. Long-term surgical outcome of masculinizing genitoplasty in large cohort of patients with disorders of sex development. J Urol. 2010 Sep;184(3):1122-7. doi: 10.1016/j.juro.2010.05.022. Epub 2010 Jul 21. PMID 20650476
- [Background] Speiser PW, Azziz R, Baskin LS, Ghizzoni L, Hensle TW, Merke DP, Meyer-Bahlburg HF, Miller WL, Montori VM, Oberfield SE, Ritzen M, White PC; Endocrine Society. Congenital adrenal hyperplasia due to steroid 21-hydroxylase deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2010 Sep;95(9):4133-60. doi: 10.1210/jc.2009-2631. PMID 20823466
- [Background] Gupta DK, Shilpa S, Amini AC, Gupta M, Aggarwal G, Deepika G, Kamlesh K. Congenital adrenal hyperplasia: long-term evaluation of feminizing genitoplasty and psychosocial aspects. Pediatr Surg Int. 2006 Nov;22(11):905-9. doi: 10.1007/s00383-006-1765-x. PMID 16947028
- [Background] Oswiecimska JM, Paradysz A, Zyczkowski M, Ziora KT, Pikiewicz-Koch A, Stojewska M, Dyduch A. Effects of feminizing surgery for ambiguous genitalia - a novel scale for evaluation of cosmetic and anatomical results. Neuro Endocrinol Lett. 2009;30(2):262-7. PMID 19675521
- [Background] Stikkelbroeck NM, Beerendonk CC, Willemsen WN, Schreuders-Bais CA, Feitz WF, Rieu PN, Hermus AR, Otten BJ. The long term outcome of feminizing genital surgery for congenital adrenal hyperplasia: anatomical, functional and cosmetic outcomes, psychosexual development, and satisfaction in adult female patients. J Pediatr Adolesc Gynecol. 2003 Oct;16(5):289-96. doi: 10.1016/s1083-3188(03)00155-4. PMID 14597017
- [Background] Crawford JM, Warne G, Grover S, Southwell BR, Hutson JM. Results from a pediatric surgical centre justify early intervention in disorders of sex development. J Pediatr Surg. 2009 Feb;44(2):413-6. doi: 10.1016/j.jpedsurg.2008.10.101. PMID 19231546
- [Background] Migeon CJ, Wisniewski AB, Gearhart JP, Meyer-Bahlburg HF, Rock JA, Brown TR, Casella SJ, Maret A, Ngai KM, Money J, Berkovitz GD. Ambiguous genitalia with perineoscrotal hypospadias in 46,XY individuals: long-term medical, surgical, and psychosexual outcome. Pediatrics. 2002 Sep;110(3):e31. doi: 10.1542/peds.110.3.e31. PMID 12205281